CLINICAL TRIAL: NCT02666183
Title: Online Information and Support for Distance Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE6Y15
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer
Keywords: cancer; caregiver; videoconferencing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Study personnel administering questionnaire and follow-up questions with participants will be blinded to the arm assignment of the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Closer (Experimental): The full intervention (Closer) is a tested intervention that uses videoconferencing technology (WebEx) for delivery and delivers the highest dose of the intervention. This arm of the intervention will deliver personalized information to the DCG (aimed at enhancing self-efficacy) and emotional support via nurse coaching as well as the opportunity for the DCG to talk with the oncologist and patient in "real time" during a minimum of four patient-oncologist office visits over a 4-month period (at least once/month). For patients who have more than one oncologist-patient meeting/month, the study will use the videoconference technology to allow the DCG to join as many of the join in as many of the oncologist-patient office visits as desired.
  Interventions: Behavioral: Video-C; Behavioral: Nurse Coaching
- Video-C Only (Active Comparator): This arm will involve the delivery of information solely via the use of videoconference technology during the patient-oncologist-DCG visit. There is always the possibility that the DCG will receive emotional support from the oncologist during the office visit (as would potentially occur during a face-to-face meeting) - but this will not be "delivered" systematically as in the Closer intervention. As with the Closer intervention, the DCG will be able to participate in the patient-oncologist visit in "real time" during a minimum of four office visits over the 4-month study period (total dose ~5 hours). The procedure for these meetings will be the same as outlined for Closer but will not involve having the nurse involved in the videoconference sessions with the oncologist, patient, and DCG.
  Interventions: Behavioral: Video-C
- Web-Only (Active Comparator): This group will be provided access to a website that will provide the following major links: a) Caregiving Resources (links to National Family Caregiver Association," etc.), b)Resources for DCGs (links to the Caregiving from a Distance," etc.), c) Cancer Information (links to National Cancer Institute, etc.). DCGs will be told that the study team will track usage of the website in order to assess which areas of the website are used most frequently. Any questions or concerns regarding use of the website can be sent online to the study's technical site, and the support staff will respond within 24 hours. As is current practice, DCGs can call an oncology nurse or oncologist to ask specific questions. Web-Only will deliver the lowest dose of the intervention.
  Interventions: Behavioral: Web-Only

INTERVENTIONS:
Behavioral: Video-C — use videoconferencing to provide personalized information aimed at enhancing self -efficacy and providing emotional support for distant caregivers of patients with advanced cancers
  Other Names: Video Conferencing
  Arms: Closer; Video-C Only
Behavioral: Nurse Coaching — structured conversations with registered nurses aimed at providing emotional support
  Arms: Closer
Behavioral: Web-Only — Access to a website with caregiving resources, resources for distant care givers, and cancer information
  Arms: Web-Only

SUMMARY:
This study seeks to test the effectiveness of two arms of an intervention that use videoconference technology for distance caregivers of patients with advanced cancer. The study is significant because the intervention will promote involvement of caregivers of patients with cancer and makes a compelling case for significance based on changing demographics and lifestyles.

DETAILED DESCRIPTION:
The primary goal of this randomized clinical trial is to compare outcomes (anxiety, distress, depression, health status) for distant care givers (DCGs) of patients with advanced cancer who are randomly assigned to either the full intervention arm (Closer), the video-only intervention arm (Video-C Only) or the control group (Web-Only). the goal is to determine which is most efficacious in improving outcomes over time for these caregivers. In addition, this study will examine the indirect effects of each arm of the intervention on DCG outcomes over time as well as explore the nature of relationships between patient and DCG distress, anxiety and depression over time.

The specific research questions include:

1. Is there a difference in DCG outcomes (anxiety, distress, depression, health status) over time between caregivers in the Closer, Video-C Only, and Web-Only groups, controlling for DCG demographic variables?
2. Are there significant indirect effects of Closer, Video-C Only, and Web-Only on DCG outcomes (anxiety, distress, depression, health status) over time, controlling for DCG demographic variables?
3. Are there significant relationships between DCG distress, anxiety, depression and health status and patient distress, anxiety and depression over time?

ELIGIBILITY:
Patient Inclusion Criteria:

* a new diagnosis (within 3 months) of advanced cancer and/or patients receiving ongoing care from a medical oncologist (solid tumors) or a new recurrence of the primary cancer in an advanced stage
* receives ongoing care from a medical oncologist at the Seidman Cancer Center
* Has English as the primary language
* Has a life expectancy of >6 months
* Provides consent for his/her own treatment and procedures
* Identifies a distant care giver (DCG) involved in his/her care, support or planning

Patient Exclusion Criteria:

* The patient sample is limited to patients with advanced cancer and/or patients receiving ongoing care from a medical oncologist because the full intervention is tailored to meet the needs of DCGs of patients with advanced cancer and/or patients receiving ongoing care from a medical oncologist

Caregiver Inclusion Criteria

* Is an adult family member (at least 18 years old) of a patient with an advanced-stage cancer
* Identifies himself/herself as a DCG for the patient
* Lives >1 hour travel time away from the patient
* Has English as his/her primary language
* Is capable of providing informed consent
* Will be able to access the internet (phone, computer, etc.)

Caregiver Exclusion Criteria

* Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Douglas, RN, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Blackstone E, Lipson AR, Douglas SL. Closer: A videoconference intervention for distance caregivers of cancer patients. Res Nurs Health. 2019 Aug;42(4):256-263. doi: 10.1002/nur.21952. Epub 2019 May 22. PMID 31119765
- [Result] Douglas SL, Mazanec P, Lipson AR, Day K, Blackstone E, Bajor DL, Saltzman J, Krishnamurthi S. Videoconference Intervention for Distance Caregivers of Patients With Cancer: A Randomized Controlled Trial. JCO Oncol Pract. 2021 Jan;17(1):e26-e35. doi: 10.1200/OP.20.00576. PMID 33434451
- [Result] Blackstone E, Douglas SL, Lipson AR. Videoconferencing Empowers Distance Caregivers to Be More Involved in Care. Oncol Nurs News. 2019 Jan-Feb;13(1):https://www.oncnursingnews.com/view/videoconferencing-empowers-distance-caregivers-to-be-more-involved-in-care. Epub 2019 Feb 8. PMID 35782672
- [Result] Douglas SL, Mazanec P, Lipson AR, Blackstone E, Day K, Bajor DL, Krishnamurthi SS. Video conference intervention for distance caregivers (DCGs) of patients with cancer: Improving psychological outcomes. Journal of Clinical Oncology. 2020; 38:15 (supplement); 12123.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closer | Video-C Only | Web-Only
Started | 137 | 141 | 119
Completed | 103 | 106 | 93
Not Completed | 34 | 35 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closer | Video-C Only | Web-Only | Total
Number analyzed (Participants) | 103 | 106 | 93 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.6) | 45.9 (12.7) | 46.8 (12.4) | 46.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 73 | 223
  Male | 28 | 31 | 20 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 1 | 7
  Not Hispanic or Latino | 81 | 86 | 73 | 240
  Unknown or Not Reported | 17 | 19 | 19 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 33 | 18 | 29 | 80
  White | 65 | 85 | 60 | 210
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 103 | 106 | 93 | 302
PROMISR SFv1.0-ED-anxiety-SF8a [Mean (Standard Deviation); unit: T-scores] | 54.66 (7.77) | 54.68 (7.14) | 56.03 (8.21) | 55.09 (7.70)
PROMISR SFv1.0-ED-depression-SF8a [Mean (Standard Deviation); unit: T-scores] | 49.64 (7.73) | 50.16 (7.92) | 52.28 (7.42) | 50.64 (7.76)
NCCN distress thermometer [Mean (Standard Deviation); unit: units on a scale] | 4.23 (2.61) | 4.00 (2.68) | 4.55 (2.39) | 4.25 (2.57)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety T-scores
Description: Compare the direct effects of Closer, Video-C Only, and Web-Only on anxiety over time, controlling for DCG demographic variables. Anxiety will be measured using the 4-item tool from the Patient Reported Outcomes measurement Information System (PROMIS). Higher scores indicate greater anxiety.
  The PROMIS Item Bank v1.0-Emotional Distress-Anxiety - Short Form 4a, a 4 item instrument, is reported as a t-score and can range from 37.1 to 83.1 with higher t-scores representing more anxiety.
  The mean and standard deviation are as follows: M=50 (SD=10).
  T-scores from 55-60 represent mild anxiety, 61-70 moderate anxiety and > 70 represent severe anxiety.
Time Frame: At enrollment to end of intervention period (4 months)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Closer | Video-C Only | Web-Only
Number analyzed (Participants) | 103 | 106 | 93
T-score | 53.14 (8.14) | 55.47 (7.67) | 56.85 (8.73)
Statistical Analysis 1: Comparison: Closer vs Video-C Only; Test type: Other; p = 0.162, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -2.251, 95% CI 2-sided [-5.051 to 0.550]
Statistical Analysis 2: Comparison: Closer vs Web-Only; Test type: Other; p = 0.007, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -3.663, 95% CI 2-sided [-6.538 to -0.789]
Statistical Analysis 3: Comparison: Video-C Only vs Web-Only; Test type: Other; p = 0.714, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -1.413, 95% CI 2-sided [-4.290 to 1.464]

2. Primary Outcome: Change in Distress Scores
Description: Compare the direct effects of Closer, Video-C Only, and Web-Only on distress over time, controlling for DCG demographic variables. Distress is conceptually defined as a negative state in which coping and adaptation processes fail to return the individual to physiological and/or psychological homeostasis. It will be measured using the National Comprehensive Cancer Network (NCCN) distress thermometer - a clinical tool currently utilized with the cancer population.
  The National Comprehensive Cancer Network Distress Thermometer is a one-item, 11-point Likert scale represented on a visual graphic of a thermometer that ranges from 0 (no distress) to 10 (extreme distress), with which patients indicate their level of distress over the course of the week prior to assessment.
  Scores range from 0 to 10 with higher scores representing higher levels of distress.
  Scores >4 indicate distress requiring further evaluation.
Time Frame: At enrollment to end of intervention period (4 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closer | Video-C Only | Web-Only
Number analyzed (Participants) | 103 | 106 | 93
score on a scale | 3.37 (2.80) | 3.89 (2.64) | 4.86 (2.66)
Statistical Analysis 1: Comparison: Closer vs Video-C Only; Test type: Other; p = 0.173, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -0.531, 95% CI 2-sided [-1.297 to 0.234]
Statistical Analysis 2: Comparison: Closer vs Web-Only; Test type: Other; p = 0.001, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -1.456, 95% CI 2-sided [-2.241 to -0.671]
Statistical Analysis 3: Comparison: Video-C Only vs Web-Only; Test type: Other; p = 0.021, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -0.925, 95% CI 2-sided [-1.711 to -0.139]

3. Primary Outcome: Change in Depression T-scores
Description: Compare the direct effects of Closer, Video-C Only, and Web-Only on depression over time, controlling for DCG demographic variables. Depression will be measured using the 4 item PROMIS Item Bank v1.0 - Emotional Distress-Depression - Short Form 4a.
  The PROMIS Item Bank v1.0 - Emotional Distress-Depression - Short Form 4a, a 4 item instrument, is reported as a t-score and can range from 38.2 to 81.3 with higher t-scores representing worse depression.
  T-scores from 55-60 represent mild depression, 61-70 moderate depression and > 70 represent severe depression.
Time Frame: At enrollment to end of intervention period (4 months)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Closer | Video-C Only | Web-Only
Number analyzed (Participants) | 103 | 106 | 93
T-score | 49.29 (8.00) | 50.72 (7.89) | 52.62 (8.75)
Statistical Analysis 1: Comparison: Closer vs Video-C Only; Test type: Other; p = 0.323, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -0.984, 95% CI 2-sided [-2.939 to 0.971]
Statistical Analysis 2: Comparison: Closer vs Web-Only; Test type: Other; p = 0.086, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -1.768, 95% CI 2-sided [-3.785 to 0.249]
Statistical Analysis 3: Comparison: Video-C Only vs Web-Only; Test type: Other; p = 0.443, ANCOVA; Covariates: DCG age, gender, race, income; Estimated marginal mean difference = -0.784, 95% CI 2-sided [-2.794 to 1.226]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout study period (6 months).
Arm/Group | Closer | Video-C Only | Web-Only
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/106 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/106 | 0/93
Other Adverse Events (participants affected / at risk) | 0/103 | 0/106 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT02666183/Prot_SAP_001.pdf